CLINICAL TRIAL: NCT06745648
Title: Effectiveness of Carotid Sinus Massage in Modified Trendelenburg Position for Acute Headache Episodes: A Pilot Study
Brief Title: Carotid Sinus Massage in Trendelenburg Position for Headache Relief
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Municipal Pedro T. Orellana (Other)
Collaborators: Duke University Medical Center, Durham, NC (Unknown)
Responsible Party: Principal Investigator, Pablo D. Anaya, MD, Principal Investigator, Hospital Municipal Pedro T. Orellana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HMPTOrellana
Record Dates: First submitted 2024-12-13; First posted 2024-12-20 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Migraine; Tension-Type Headache
Keywords: Carotid Sinus Massage; Trendelenburg; Autonomic Nervous System
MeSH Terms: conditions — Migraine Disorders; Tension-Type Headache

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of two parallel arms: (1) real carotid sinus massage in the Trendelenburg position (CSM+T), or (2) a sham neck massage in the same position. The primary outcome will compare immediate post-intervention headache intensity between groups.
Who Masked: Participant
Masking Description: In this single-blinded design, the patients do not know whether they are receiving the real CSM+T or the sham intervention, ensuring unbiased reporting of pain outcomes. However, it is not possible to double-blind (i.e., also blind the healthcare providers) because the clinicians administering CSM+T or the sham procedure must be aware of which maneuver they are performing, making true double-blinding impractical in this hands-on intervention study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A - Carotid Sinus Massage + Trendelenburg (CSM+T) (Experimental): Participants will receive carotid sinus massage (CSM) while positioned in a 10-15° Trendelenburg position. The massage is applied to the carotid sinus area for approximately 5 seconds and may be repeated up to three times, separated by one-minute intervals. Pain intensity and vital signs are assessed before and after the intervention.
  Interventions: Procedure: Arm A - Carotid Sinus Massage + Trendelenburg (CSM+T)
- Arm B - Sham CSM+T (Sham Comparator): In the control group, patients will be placed in the supine position. Then, a sham neck massage will be performed by lightly touching the skin in a circular motion away from the carotid sinus, for the same duration and intervals as in the experimental procedure. This sham approach will ensure that any observed effects are attributable to carotid sinus stimulation rather than mere tactile stimulation of the neck.
  Participants who do not report pain relief after the sham procedure will be offered rescue therapy, which may include the real CSM+Trendelenburg intervention or pharmacologic treatment, as clinically appropriate. The rescue response will be recorded for secondary analysis.
  Interventions: Procedure: Arm B - Sham CSM+T

INTERVENTIONS:
Procedure: Arm A - Carotid Sinus Massage + Trendelenburg (CSM+T) — Manual stimulation of the carotid sinus area combined with head-down tilt positioning to activate baroreceptors for headache relief.
  Arms: Arm A - Carotid Sinus Massage + Trendelenburg (CSM+T)
Procedure: Arm B - Sham CSM+T — Light neck contact, avoiding carotid sinus pressure, paired with identical body positioning to mimic the experimental intervention.
  Arms: Arm B - Sham CSM+T

SUMMARY:
Headaches significantly impact patients' quality of life, with tension-type headaches and migraines being among the most prevalent types. There is growing evidence suggesting that blood pressure regulation and baroreceptor activity play a role in headache pathophysiology. Carotid sinus massage (CSM), particularly when combined with the modified Trendelenburg position, may modulate autonomic nervous system activity to relieve headache symptoms.

An initial open-label pilot study (n = 17) was completed, and the results were published in a preprint server for health sciences, the Medical Research Archive (medRxiv), demonstrating the feasibility, safety, and promising preliminary efficacy of CSM+T. Based on these findings, a follow-up randomized, sham-controlled, parallel-arm trial will further evaluate the efficacy of the treatment.

DETAILED DESCRIPTION:
This protocol includes two study phases:

1. Pilot Phase (Completed): A single-arm, open-label pilot study was conducted in 17 participants to assess the feasibility and safety of CSM+T for the relief of headaches. Results have been published in medRxiv and support continued investigation.
2. Parallel-Arm Phase (Planned): A randomized, sham-controlled, parallel-arm clinical trial will now be implemented to evaluate efficacy. This phase will enroll 18 participants (9 per arm) to detect a clinically meaningful difference in headache relief with 80% power (α = 0.05, two-sided), accounting for potential attrition.

ELIGIBILITY:
INCLUSION CRITERIA:

* Participants must be at least 16 years of age.
* Must have a diagnosis of one of the following, according to the International Classification of Headache Disorders (ICHD-3):

  * Migraine
  * Tension-type headache
  * Mixed headache
* The headache episode must have started within the past 24 hours.

EXCLUSION CRITERIA:

* Any contraindication to carotid sinus massage, including:

  * Carotid bruits
  * Recent myocardial infarction
  * History of stroke
  * Known or suspected carotid artery stenosis
* Any contraindication to the Trendelenburg position, including:

  * Increased intracranial pressure
  * Respiratory distress
  * Congestive heart failure
  * History of syncope
  * History of cardiac arrhythmias

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-12-21 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in headache pain intensity | Baseline to 15 minutes post-intervention
  Change in self-reported pain intensity using a 10-point Visual Analog Scale (VAS)

SECONDARY OUTCOMES:
Change in blood pressure | Baseline to 15 minutes post-intervention
  Difference in systolic and diastolic blood pressure (mmHg) from baseline to 15 minutes after the intervention.
Change in heart rate | Baseline to 15 minutes post-intervention
  Difference in heart rate (beats per minute) measured before and after the intervention to assess autonomic or cardiovascular effects of the treatment.
Change in oxygen saturation | Baseline to 15 minutes post-intervention
  Difference in peripheral oxygen saturation (SpO₂, %) measured by pulse oximetry before and after the intervention.
Percentage of participants with complete pain relief (VAS = 0) | 15 minutes post-intervention
  Proportion of participants reporting a Visual Analog Scale (VAS) pain score of 0-indicating complete headache relief-15 minutes after the intervention.
  VAS scores range from 0 (no pain) to 10 (worst possible pain)
Headache recurrence rate | 24 hours post-intervention
  Proportion of participants who experience recurrence of headache symptoms within 24 hours following the intervention.
Incidence of adverse events | Up to 24 hours post-intervention
  Number and type of adverse events reported within 24 hours of the intervention, including any hemodynamic instability, discomfort, or other complications.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo D Anaya, MD, Principal Investigator — Hospital Municipal Pedro T. Orellana; Heberto J Suarez-Roca, MD, PhD, Study Director — Dule University Medical Center, Dept. of Anesthesiology, Center for Translational Pain Medicine
Locations (1):
- Hospital Pedro T.Orellana, Trenque Lauquen, Trenque Lauquen, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to study outcomes will be shared, including pain scores, physiological measurements (such as heart rate, blood pressure, and oxygen saturation), and adverse event reports. Data will be made available upon reasonable request after publication of the primary results.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: IPD will be made available beginning 6 months after publication of the primary results and will remain available for a minimum of 5 years thereafter.
Access Criteria: Qualified researchers may request access to the data by submitting a data use proposal, which should include a brief description of the study objectives and statistical plan. Requests will be reviewed by the study investigators or a designated data access committee. Data will be shared via secure transfer methods, subject to a data use agreement, to ensure participant confidentiality.